CLINICAL TRIAL: NCT01902940
Title: Retrospective Cohort Study Assessing the Natural Course in Congenital Cataract Facial Dysmorphism Neuropathy Syndrome (CCFDN) and Sporadic and Hereditary Inclusion Body Myopathies (IBM)
Brief Title: Natural History in CCFDN and IBM Syndromes
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Maggie Walter, Professor, MD, MA, Ludwig-Maximilians - University of Munich
Other Study IDs: CCFDN-IBM-2013; CCFDN-IBM-2013 (Other: Friedrich-Baur-Institute)
Record Dates: First submitted 2013-07-03; First posted 2013-07-18 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Inclusion Body Myositis, Sporadic; Inclusion Body Myopathy, Autosomal-recessive; Inclusion Body Myopathy, Autosomal-dominant; Congenital Cataracts, Facial Dysmorphism, And Neuropathy
MeSH Terms: conditions — Myositis, Inclusion Body; Distal myopathy, Nonaka type; Inclusion body myopathy, autosomal dominant; Congenital Cataracts, Facial Dysmorphism, And Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Natural History: Assessment of natural history in IBM and CCFDN
  Interventions: Other: Natural History

INTERVENTIONS:
Other: Natural History — Assessment of natural history in IBM and CCFDN

SUMMARY:
So far, only limited data is available regarding the natural course in Congenital Cataract Facial Dysmorphism Neuropathy Syndrome (CCFDN) and sporadic and hereditary inclusion body myopathies (IBM). Several criteria and outcome measures have led to contradicting results. The investigators want to retrospectively assess the natural course of the disease in CCFDN and IBM patients according to the data recorded during clinical routine visits.

DETAILED DESCRIPTION:
We wanted to assess the natural course in Congenital Cataract Facial Dysmorphism Neuropathy Syndrome (CCFDN) and sporadic and hereditary inclusion body myopathies (IBM) over 10 years to gain new insights in both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or genetic diagnosis of Congenital Cataract Facial Dysmorphism Neuropathy Syndrome (CCFDN) and sporadic and hereditary inclusion body myopathies (IBM)

Exclusion Criteria:

* Additional neuromuscular diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CCFDN and IBM
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Strength assessed by Medical Research Council (MRC) | 6-months intervals
  Retrospective

CONTACTS AND LOCATIONS:
Overall Officials: Maggie C Walter, MD, MA, Study Chair — Friedrich-Baur-Institute, Dept. of Neurology
Locations (1):
- Friedrich-Baur-Institut, Ludwig-Maximilians-University of Munich, Munich, Bavaria, Germany